CLINICAL TRIAL: NCT05200260
Title: A Prospective, Multicenter, Randomized Phase II Trial on Optimal Timing of Surgery Combined With Maintenance Targeted Therapy in the Treatment of Advanced Ovarian Cancer
Brief Title: Surgery Combined With Maintenance Targeted Therapy in the Treatment of Advanced Ovarian Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Gynecologic Oncology Group (Other Government)
Collaborators: Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAT-1
Record Dates: First submitted 2022-01-17; First posted 2022-01-20 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2024-11

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Primary Peritoneal Carcinoma
Keywords: Ovarian Cancer; Primary Debulking Surgery; Neoadjuvant chemotherapy; Poly-adenosine Ribose Phosphate Inhbitors (PARPi); Bevacizumab
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms | interventions — Neoadjuvant Therapy; Poly(ADP-ribose) Polymerase Inhibitors; olaparib; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Upfront cytoreductive surgery with maintenance therapy (Experimental): Primary debulking surgery with a maximal cytoreduction of complete gross resection within 3 weeks after biopsy, followed by at least 6 cycles of adjuvant chemotherapy and maintenance therapy for patients with CR/PR after platinum-based therapy (patients with or without BRCA mutation will be maintained by PARPi or Bevacizumab respectively ).
  Interventions: Procedure: Primary debulking surgery; Drug: PARP inhibitor; Drug: Bevacizumab
- Neoadjuvant chemotherapy with maintenance therapy (Active Comparator): Neoadjuvant chemotherapy with 3 cycles of chemotherapy, then followed by interval debulking surgery. The maximal time interval between course 3 chemotherapy and IDS is 6 weeks. And then 3 cycles of adjuvant chemotherapy and maintenance therapy for patients with CR/PR after platinum-based therapy (patients with or without BRCA mutation will be maintained by PARPi or Bevacizumab respectively ).
  Interventions: Procedure: Neoadjuvant chemotherapy; Drug: PARP inhibitor; Drug: Bevacizumab

INTERVENTIONS:
Procedure: Primary debulking surgery — Primary debulking surgery with a maximum cytoreduction, then followed by 6 cycles of Paclitaxel 175mg/m2 or Docetaxel 60-75 mg/m2 plus Carboplatin AUC (area under the curve) 5.
  Other Names: PDS
  Arms: Upfront cytoreductive surgery with maintenance therapy
Procedure: Neoadjuvant chemotherapy — 3 cycles of Paclitaxel 175mg/m2 or Docetaxel 60-75 mg/m2 plus Carboplatin AUC (area under the curve) 5, Interval debulking surgery with a maximal cytoreduction of complete gross resection, then followed by another 3 cycles of chemotherapy.
  Other Names: Neoadjuvant chemotherapy followed by interval debulking surgery, NACT-IDS
  Arms: Neoadjuvant chemotherapy with maintenance therapy
Drug: PARP inhibitor — For patients with BRCA mutated, maintenance therapy of PARP inhibitors following CR/PR after first-line chemotherapy. In this trial, Olaparib 300mg p.o. twice daily is suggested after the front-line therapy.
  Other Names: Olaparib
Drug: Bevacizumab — For patients without BRCA mutated, maintenance therapy of Bevacizumab following CR/PR after first-line chemotherapy. In this trial, Bevacizumab 7.5mg per kilogram intravenous once every 3 weeks is suggested after the front-line therapy.

SUMMARY:
Optimal Timing of Surgery combined with Maintenance Therapy in the Front-line Treatment of Advanced Ovarian Cancer

DETAILED DESCRIPTION:
The purpose of this trial is to answer the fundamental question 'The Optimal Timing of Surgery' combined with Bevacizumab or Poly-adenosine Ribose Phosphate Inhbitors (PARPi), in the circumstance of primarily diagnosed advanced epithelial ovarian cancer, fallopian tube cancer and primary peritoneal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Females aged ≥ 18 years.
* Pathologic confirmed stage IIIC and IV epithelial ovarian cancer, fallopian tube cancer or primary peritoneal carcinoma
* Low, Middle tumor burden and high tumor burden with cPCI score ≤ 12 based on pre-operative CT or PET/CT examination
* Complete cytoreduction can be achieved based on CT or PET/CT examination
* Patients must agree to undergo BRCA (breast cancer gene) and HRD (homologous recombination deficiency) testing
* Performance status (ECOG 0-2)
* Adequate bone marrow, renal and hepatic function to receive chemotherapy and subsequent surgery:

  1. white blood cells >3,000/µL, absolute neutrophil count ≥1,500/µL, platelets ≥100,000/µL, hemoglobin ≥9 g/dL,
  2. serum creatinine <1.25 x upper normal limit (UNL) or creatinine clearance ≥60 mL/min according to Cockroft-Gault formula or to local lab measurement,
  3. serum bilirubin <1.25 x UNL, AST(SGOT) and ALT(SGPT) <2.5 x UNL.
* Comply with the study protocol and follow-up.
* Patients who have given their written informed consent.

Exclusion Criteria:

* Non-epithelial ovarian malignancies and borderline tumors
* Low grade ovarian cancer
* Mucinous ovarian cancer
* Complete cytoreduction cannot be achieved according to preoperative evaluation, including pulmonary and hepatic parenchymal metastases, unresectable extensive pleural metastases, multiple thoracic lymph nodes metastases, brain or bone metastases
* Patient has a known hypersensitivity to the components of olaparib/bevacizumab or its excipients
* Synchronous or metachronous (within 5 years) malignancy other than carcinoma in situ, thyroid carcinoma, or breast carcinoma (without any signs of relapse or activity, early-stage).
* Any other concurrent medical conditions contraindicating surgery or chemotherapy that could compromise adherence to the protocol.
* Other conditions, such as religious, psychological, and other factors, that could interfere with the provision of informed consent, compliance to study procedures, or follow-up.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 220 (Estimated)
Dates: Start 2022-07-13 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
3-year overall survival | Participants will be followed for at least 3 years after randomization
  The proportion of patients alive at 3 years after entry into the study

SECONDARY OUTCOMES:
Overall survival | Participants will be followed for at least 3 years after randomization
  Time from entry into the study to any cause of death
Progression-free survival | Participants will be followed for at least 3 years after randomization
  Time from entry into the study to the diagnosis of the first progression or recurrence or death, whichever occurs first
Post-operative complications | Participants will be followed up to 3 months after randomization
  The surgical complications will be evaluated at 30-day, 60-day, 90-day after upfront cytoreductive surgery or interval debulking surgery
Quality of life assessments | Participants will be followed for at least 3 years after randomization
  QLQ-C30, FACT-Q (baseline; 6 months, 12 months, 24 months and 36 months after randomization)
Accumulated treatment-free survival | Participants will be followed for at least 3 years or death after randomization
  Time from the date of randomization to death from any reason, minus the total treatment time of surgery and chemotherapy after randomization (regardless of targeted therapy)
TFST | Participants will be followed for at least 3 years or death after randomization
  Time from the date of randomization until the starting date of the first subsequent anticancer therapy or death, whichever occurred first, whichever occurred first
TSST | Participants will be followed for at least 3 years or death after randomization
  Time from the date of randomization until the starting date of the second subsequent anticancer therapy or death, whichever occurred first
The pattern of the first relapse | Participants will be followed for at least 3 years or death after randomization
  The number and sites of the first relapse, including pelvic, abdominal, retroperitoneal lymph nodes, distant metastases and ascites will be compared between the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Libing Xiang, Study Chair — Fudan University
Locations (9):
- China (9):
  - The First People's Hospital of Foshan, Foshan
  - Sun Yet-Sen University Cancer Center, Guangzhou
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - The First Affiliated Hospital of University of Science and Technology of China, Hefei
  - Fudan University Cancer Hospital, Shanghai
  - Obstetrics and Gynecology Hospital of Fundan University, Shanghai
  - Xinhua Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai
  - Zhongshan Hospital, Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: No